CLINICAL TRIAL: NCT00857922
Title: Neurosciences Research Repository
Acronym: NRR
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Georgene Hergenroeder, Study Director, PI, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-08-0413
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Neurological Conditions
Keywords: Neurological; Neurosurgical
MeSH Terms: conditions — Neurologic Manifestations | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, white cells, saliva, tissue, CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurosurgical patient: Neurosurgical patient of the Mischer Neuroscience Institute, 18 years and over
  Interventions: Other: tissue and data repository
- Family members: Family members of specific vascular, trauma, brain tumor and functional disorder cohorts
  Interventions: Other: tissue and data repository

INTERVENTIONS:
Other: tissue and data repository — Tissue and data will be maintained in a repository for study from consenting subjects.

SUMMARY:
In order to expand neuroscience research and move laboratory advances to patients, there is a need to integrate reliable clinical data with biologic information from patient tissue specimens. The Neuroscience Research Repository (NRR) seeks to meet this need. The NRR is a prospective database and sample bank created to collect information and samples for current and future neuroscience research. The objective of this NRR is to develop a data and sample repository for study of neurological conditions. A repository utilizing standardized electronic health data and samples collected in a uniform manner serves to foster the ability to perform research on current and future projects. Samples and data for clinical, genomic and proteomic analysis will be provided to optimize their value for neuroscience research.

The NRR will enroll patients and collect clinically recorded longitudinal data for as long as they are followed by the Neurosurgery service and up to an additional 5 years after being released from care. Patients will be enrolled on admission to the service and samples will be taken at three time points: Time One, within 24 hours of event (preferably first blood draw); Time Two, within 48 hours of event; and Time Three, time of any residual tissue availability. Family members of select groups of patients will also be approached for enrollment.

Samples and data will be labeled with a study code to maintain confidentiality. Samples and data will be maintained in secure, limited access environments with back-up/redundancy procedures in place. Sample inventory will be maintained with a bar-coding system. A duty to warn clause will be included in the consent as will the determination of willingness to be re-contacted for future research. Time of sample acquisition to time of sample processing will be documented for quality control purposes. Freezers will be monitored for temperature stability. Recipient investigators will be requested to provide feedback on sample quality. Samples will be distributed to neuroscience investigators after approval from the Neurosurgery Scientific Review Committee - Dissemination Review Committee and the Committee for the Protection of Human Subjects (CPHS).

ELIGIBILITY:
Inclusion Criteria:

1. Neurosurgical patient (primary or consulting); patients<18 includes residual tissue only, no blood samples.
2. Family members of specific vascular, trauma, brain tumor and functional disorder cohorts (will be identified in future addendums to this repository)

Exclusion Criteria:

1. Inability to obtain informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the Neurosurgery service (Mischer Neuroscience Institute/UT Department of Neurosurgery or Neurosurgical Critical Care service) are eligible for this study. Family members of those with select conditions will be approached for enrollment at a future date.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Discharge status | hospital discharge
  Standardized functional outcome score

CONTACTS AND LOCATIONS:
Overall Officials: Georgene W Hergenroeder, PhD, Principal Investigator — McGovern Medical School at UTHealth
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States